CLINICAL TRIAL: NCT04967391
Title: The Role Of Tumescence In Split Thickness Skin Grafting For Reconstruction Of Head And Neck Cancer Resection
Brief Title: Tumescence in HNC Skin Graft Reconstruction
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1777948
Record Dates: First submitted 2021-06-21; First posted 2021-07-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer; Surgery--Complications; Graft Failure
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: saline vs saline with epinephrine
Who Masked: Participant, Investigator
Masking Description: Participants will be masked to the randomization group. Investigators that will be reviewing the graft images will also be masked to the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tumescence During STSG Harvest (Experimental): Prior to the split thickness skin graft (STSG) harvest, the tumescence technique will injection of 100-150 mL normal saline with 1:500,000 epinephrine injected into a deep dermal thigh tissue plane with 18-gauge spinal needle on a 60 mL syringe.
  Interventions: Procedure: Tumescence During STSG Harvest
- No Intervention (No Intervention): Patients randomized to "no tumescence" will have their free flap donor site reconstructed with a split thickness skin graft (STSG) harvested at 0.0175 inches using the dermatome to obtain a graft from the thigh.

INTERVENTIONS:
Procedure: Tumescence During STSG Harvest — Tumescence injections performed prior to STSG harvest
  Arms: Tumescence During STSG Harvest

SUMMARY:
Our primary objective is to determine if the use of tumescence has a meaningful effect on STSG uptake at the recipient site. This is an important outcome because poor graft uptake results in the need for prolonged local wound care, additional clinic visits for patients and increased risk of infection. A prospective, randomized comparison of the tumescence to our current standard of care will allow us to definitively evaluate any benefits to this technique.

Tumescence is commonly used in the treatment of burn patients to minimize blood loss during both tangential excision of eschar and during harvest of split-thickness grafts for reconstruction. This is considered the standard of care in burn surgery as using tumescence has been clearly demonstrated to reduce intraoperative blood loss during harvest of large skin grafts and excision of large burns when compared with the application of topical epinephrine as was the historic standard practice.4-6 Tumescence also creates a firm and uniform surface from which to harvest the skin graft, which the investigators believe may improve the quality of harvest and rate of skin graft take.

DETAILED DESCRIPTION:
Multimodal treatment for head and neck cancer often includes surgical resection. Large tumors leave behind large anatomical defects when resected, which require reconstruction to rehabilitate form and function after ablative surgery. Two commonly used reconstructive options in reconstructive surgery are the radial forearm free flap and the fibula free flap. These in turn leave cutaneous defects at the donor site which must be reconstructed to protect the underlying soft tissues, muscles, and tendons exposed as a result of their harvest. This is effectively accomplished with a split thickness skin graft harvested from the thigh, which generally results in excellent coverage of the free flap donor site and minimal skin graft donor site morbidity. 1-3 Using a free flap for reconstruction following surgical tumor ablation often leaves behind a donor site that cannot be closed primarily and at our institution these defects are reconstructed using split-thickness skin grafts (STSG) harvested from the thigh. This creates an additional wound that must be carefully monitored, as poor skin graft take or failure can result in exposed muscle or tendon at the donor site. While many of these wound-healing complications can be treated with simple dressings, this can create added stress, another site of potential infection, and delayed healing and return to function.1-3 Tumescence of the skin graft harvest site involves a deep dermal infiltration of normal saline with epinephrine to the thigh prior to skin graft harvest. This has been demonstrated to minimize intraoperative blood loss4-6 and is routinely utilized in burn surgery where extensive skin grafting is often required.

The effect of tumescence on skin graft quality and take has not been evaluated. Anecdotally, it is our impression that this procedure may yield a lower graft failure rate thereby decreasing post-operative extremity immobility, risk of infection and wound care requirements.2 In this study, the investigators plan to compare the quality and take of split thickness skin grafts harvested with and without tumescence. Our results will have important implications for how split thickness skin grafting is performed in head and neck reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria Patients must meet all of the following criteria to be eligible for study entry.

1. Ability to adhere to the study visit schedule and other protocol requirements.
2. Men and women ≥18 years of age.
3. Life expectancy ≥ 3 months.
4. Planned surgery for head and neck cancer ablation requiring split-thickness skin grafting for reconstruction of free flap donor sites from the forearm and fibula.

Exclusion Criteria Patients who meet any of the following criteria will be excluded from study entry.

1. Pregnant or lactating women.
2. History of prior radiation.
3. Any significant medical condition which, in the opinion of the investigator, will not be appropriate for the study.
4. Severe infection that in the opinion of the investigator would interfere with patient safety or compliance on trial within 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of graft uptake | One Month Post-op
  To assess the use of tumescence during STSG harvest affect graft take at the recipient site as measured by percentage of graft uptake as measured using ImageJ (open source software available from NIH) at one month post-operatively

SECONDARY OUTCOMES:
The Occurence of Graft Locations | One Month Post-op
  To determine whether the location of the graft (radial forearm v fibula) affects the graft take.
Size of skin graft | One Month Post-op
  To determine whether the size of the recipient site defect affect graft take.
Incidence of Smoking Status Comorbidity | One Month Post-op
  To evaluate if comorbidities including smoking status affect skin graft take.
Incidence of Diabetes Comorbidity | One Month Post-op
  To evaluate if comorbidities including Diabetes affect skin graft take.
Incidence of BMI Comorbidity | One Month Post-op
  To evaluate if comorbidities including BMI affect skin graft take.
Incidence of Peripheral Arterial Disease Comorbidity | One Month Post-op
  To evaluate if comorbidities including Peripheral Arterial Disease affect skin graft take.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.